CLINICAL TRIAL: NCT02921880
Title: Does Cardiac REhabilitation Improve Functional, Independence, Frailty and Emotional outCOmes Following Trans Catheter Aortic ValvE Replacement?
Acronym: RECOVER-TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16/OO/0687
Record Dates: First submitted 2016-09-28; First posted 2016-10-03 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiac Rehabilitation (Experimental): Patients will return to the out-patient clinic at 4 weeks post - TAVR and research consent will be re-affirmed. Patients will be randomised to receive a programme of cardiac rehabilitation or routine care at this point. Patients randomised to receive cardiac rehabilitation will meet the cardiac rehab team and undergo baseline assessment for the programme. This involves recording height, weight, blood pressure, oxygen saturation and heart rate and rhythm. An individualised programme will be established to meet the needs of each patient. The patients will undergo a 6 week programme of cardiac rehab. Patients who are not allocated to the intervention group will not receive a cardiac programme and will have access to the TAVR nurse specialist team as would be usual care.
  Interventions: Other: Cardiac Rehabilitation
- Standard of care (No Intervention): 15 patients will be randomised to receive a programme of cardiac rehabilitation, and 15 patients will receive standard of care which does not include a routine rehabilitation programme.

INTERVENTIONS:
Other: Cardiac Rehabilitation
  Arms: Cardiac Rehabilitation

SUMMARY:
The aim of this pilot study is to assess function, independence, frailty and emotional status in 30 patients who have been accepted for TAVI. All patients will attend clinic for review at 4 weeks post implant and at that stage, 15 patients will be randomised to undertake a cardiac rehabilitation programme and the remaining 15 patients will receive standard of care. All patients will return to clinic at 3 months and 6 months post implant and undertake the functional, independence, frailty and emotional testing again.

DETAILED DESCRIPTION:
BACKGROUND

Aortic stenosis is the most common form of valvular heart disease in the elderly and is associated with high morbidity and mortality once cardiac symptoms develop (1). In patients who are at high risk for serious complications during or after surgery, Transcatheter Aortic Valve Implantation (TAVI) has been shown to result in reductions in mortality and improvement in quality of life compared with medical therapy (2, 3).

Due to the ageing and increasingly complex nature of patients with aortic stenosis, frailty and functional assessment has become a high-priority theme within patient management. Frailty is a term widely used to describe a multidimensional syndrome of loss of reserves (energy, physical ability, cognition, health) that gives rise to vulnerability. Several publications deal with the impact of frailty on mortality and morbidity in the elderly population. Functional status is evaluated by the ability to undertake Activities of Daily Living (ADL) and it has been demonstrated that frailty and the onset of dependence in ADL are strongly associated.

4.2 PRE-CLINICAL DATA/CLINICAL DATA

Cardiac rehabilitation is a complex intervention offered to patients with heart disease and includes components of health education, advice on cardiovascular risk reduction, physical activity and stress management. Cardiac rehabilitation and physical activity are recommended treatments after cardiac valve surgery and positively improves morbidity, exercise capacity and quality of life or emotional well-being. The National Institute for Healthcare Excellence and The Department of Health and wider European guidelines agree that patients who have received heart valve replacements will benefit from cardiac rehabilitation.

4.3 STUDY RATIONALE AND RISK/BENEFIT ANALYSIS

A literature search has not revealed any publications which specifically outline the impact of receiving a programme of cardiac rehabilitation, following TAVR and this study aims to address that question. The ethical dilemma of conducting research in elderly patients who have undergone TAVR can be associated with clinical trials in other elderly populations. The dilemma consists of the need to develop new and better treatment options for a particular group of patients whilst protecting the patient from harm. We anticipate that this study will allow us to understand the feasibility of undertaking this study in a group of patients who have agreed to participate in a research study prior to the TAVR procedure. The pilot study will help us to understand the logistics of providing a cardiac rehabilitation programme for patients and the data we generate will allow us to understand if there are any benefits related to functional, independence, frailty and emotional domains for this patient group. The outcomes from this pilot study may allow us to plan future studies with the aim of developing appropriate guidelines related to the provision of cardiac rehabilitation for this patient group.

4.4 MANAGEMENT OF POTENTIAL STUDY RISKS

Patients who are eligible for TAVR, as determined by the multi-disciplinary team, will be seen in the out-patient clinic or in-patient area by the Research Nurse Manager or delegated research nurse. Full informed consent will be obtained before any research intervention is undertaken. Functional, independence, frailty and emotional assessment will include 6 minute walk teat, 4m gait speed walk, hand grip strength, questionnaires and cognitive assessment.

Patients will undergo TAVR as per routine practice and they will be discharged when safe to do so. The research nurse team will collect clinical data during the admission. All patients will attend clinic for review at 4 weeks post implant, research consent will be reaffirmed and the patients will be randomised to receive a cardiac rehabilitation programme or standard of care.

A personalised programme of cardiac rehabilitation will be developed by expert physiotherapists. Patients in the cardiac rehab group will be assessed for the cardiac rehabilitation prior to any intervention taking place. Patients are monitored during exercise and full emergency equipment is available should there be an emergency.

Patients who are in the standard of care group will have access to the TAVR nurse specialist as well as the designated Consultant and research nurse team to ask any advice at any time.

ELIGIBILITY:
Inclusion Criteria:

* Severe symptomatic aortic stenosis accepted for Trans Catheter Aortic Valve Replacement
* Age ≥75 years;
* Participant able and willing to give written informed consent;
* Participant able (in the Investigator's opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Subjects may not enter the study if ANY of the following apply:
* Intervention deemed inappropriate due to co-morbidity or frailty;
* Life expectancy less than one year due to co-morbidity;
* Previous AVR or TAVI;
* Predominant aortic regurgitation (AR).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients willing to undertake cardiac rehabilitation following TAVR. | 6 months

SECONDARY OUTCOMES:
Functional capacity by 4 metre gait speed. | 6 months
  Measured at baseline, 6 weeks, 3 months and 6 months.
Frailty assessment via the FRIED criteria. | 6 months
  Measured at baseline, 6 weeks, 3 months and 6 months.
Hospital Anxiety and Depression score | 6 months
  Measured at baseline, 6 weeks, 3 months and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, Uxbridge, Middlesex, United Kingdom

REFERENCES:
- [Background] Bonow RO, Carabello BA, Chatterjee K, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2008 focused update incorporated into the ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to revise the 1998 guidelines for the management of patients with valvular heart disease). Endorsed by the Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2008 Sep 23;52(13):e1-142. doi: 10.1016/j.jacc.2008.05.007. No abstract available. PMID 18848134
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Reynolds MR, Magnuson EA, Lei Y, Leon MB, Smith CR, Svensson LG, Webb JG, Babaliaros VC, Bowers BS, Fearon WF, Herrmann HC, Kapadia S, Kodali SK, Makkar RR, Pichard AD, Cohen DJ; Placement of Aortic Transcatheter Valves (PARTNER) Investigators. Health-related quality of life after transcatheter aortic valve replacement in inoperable patients with severe aortic stenosis. Circulation. 2011 Nov 1;124(18):1964-72. doi: 10.1161/CIRCULATIONAHA.111.040022. Epub 2011 Oct 3. PMID 21969017
- [Derived] Rogers P, Al-Aidrous S, Banya W, Haley SR, Mittal T, Kabir T, Panoulas V, Raja S, Bhudia S, Probert H, Prendergast C, Spence MS, Davies S, Moat N, Taylor RS, Dalby M. Cardiac rehabilitation to improve health-related quality of life following trans-catheter aortic valve implantation: a randomised controlled feasibility study: RECOVER-TAVI Pilot, ORCA 4, For the Optimal Restoration of Cardiac Activity Group. Pilot Feasibility Stud. 2018 Dec 13;4:185. doi: 10.1186/s40814-018-0363-8. eCollection 2018. PMID 30564436